CLINICAL TRIAL: NCT01056250
Title: Performing Cholangiography During SILS Cholecystectomy: is it Feasible?
Brief Title: SILS Cholecystectomy: Cholangiography of the Biliary Tract
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St John of God Hospital, Vienna (Other)
Responsible Party: Bernhard Dauser, MD, St John of God Hospital, Vienna
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT3; SJOG 3 (Other: Ethikkommission)
Record Dates: First submitted 2010-01-24; First posted 2010-01-26 (Estimated); Last update posted 2011-05-10 (Estimated); Status verified 2010-07

CONDITIONS: Cholecystolithiasis
Keywords: cholelithiasis
MeSH Terms: conditions — Cholecystolithiasis; Cholelithiasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SILS cholangiography (Other): Performing cholangiography in all patients undergoing SILS cholecystectomy.
  Interventions: Procedure: SILS cholangiography

INTERVENTIONS:
Procedure: SILS cholangiography — intraoperative
  Other Names: LESS; E-NOTES

SUMMARY:
Single Incision Laparoscopic Surgery (SILS) can be performed for different standard operations such as appendectomy and cholecystectomy. During laparoscopic cholecystectomy sometimes a cholangiography (marking the biliary tract with contrast agent) is necessary to identify and preserve relevant structures. The investigators want to evaluate feasibility of performing cholangiography during SILS cholecystectomy.

ELIGIBILITY:
Inclusion Criteria:

* cholecystolithiasis

Exclusion Criteria:

* acute cholecystitis

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2009-09; Primary Completion 2010-11 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Feasibility of cholangiography during SILS cholecystectomy | at operation

SECONDARY OUTCOMES:
biliary tract injury | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bernhard Dauser, MD, Principal Investigator — St John of God Hospital, Vienna
Locations (1):
- St John of God Hospital, Vienna, Vienna, Austria